CLINICAL TRIAL: NCT00274846
Title: Allogeneic Natural Killer Cells in Patients With Relapsed Acute Myelogenous Leukemia
Brief Title: Donor Peripheral Stem Cell Transplant in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000450852; UMN-2004LS073 (Other: Clinical Trials Office, University of Minnesota); UMN-MT2004-25 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — aldesleukin; Interleukin-2; Lymphocyte Count; Cyclophosphamide; fludarabine phosphate; IL32 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intent-to-Treat (Experimental): All patients treated with natural killer (NK) cells (at a dose of 1.5-8 x 10^7/kg.)
  Interventions: Biological: aldesleukin; Biological: therapeutic allogeneic lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: in vitro treated peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: aldesleukin — 10 million units three times a week for a total of 6 doses. For any subject less than 45 kilograms the IL-2 will be given at 5 million units per meter squared three times weekly for a total of 6 doses
  Other Names: IL-2
Biological: therapeutic allogeneic lymphocytes — Cells infused per kg. 1.5-8.0 x 10^7/kg Total cells infused(for 70 kg. adult) 1.05 - 5.6 x 10^9
  Other Names: lymphocytes
Drug: cyclophosphamide — Days -5 and -4: 60 mg/kg
  Other Names: Cytoxan
Drug: fludarabine phosphate — Days -5 through -2: 25 mg/m^2
  Other Names: Fludara
Procedure: in vitro treated peripheral blood stem cell transplantation — Day 0 infuse natural killer cells
  Other Names: Natural Killer Cells

SUMMARY:
RATIONALE: Giving chemotherapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells and natural killer (NK) cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This clinical trial is studying how well a peripheral stem cell transplant using NK cells from a donor works in treating patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the in vivo expansion of natural killer (NK) cells 14 days after treatment with allogeneic NK cell-enriched peripheral blood stem cell transplantation in patients with relapsed acute myeloid leukemia.

Secondary

* Determine the response rate, in terms of complete remission, in patients treated with this regimen.
* Correlate complete remission rate with NK cell expansion, interleukin-15 levels, and donor/recipient killer immunoglobulin receptor (KIR) ligand matching status in patients treated with this regimen.
* Determine the overall and progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label study.

* Induction therapy: Patients receive fludarabine IV on days -6 to -2 and cyclophosphamide IV on day -5 or on days -5 and -4.
* Allogeneic natural killer (NK) cell-enriched peripheral blood stem cell transplantation: Patients receive allogeneic NK cell-enriched peripheral blood stem cells IV over 15-60 minutes on day 0. Patients also receive interleukin-2 subcutaneously beginning on day 0 and continuing 3 times a week for up to 2 weeks.

After completion of study treatment, patients are followed periodically for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) meeting 1 of the following criteria:

  * Primary refractory disease (no complete response [CR] after ≥ 2 induction therapies)
  * Relapsed disease not in CR after ≥ 1 course of standard reinduction therapy
  * Secondary AML from myelodysplastic syndromes
  * Disease relapsed ≥ 2 months after transplant and no option of donor lymphocyte infusions (e.g., recipients of autologous or umbilical cord blood transplants)
  * Chronic myelogenous leukemia with myeloid blast crisis not in second chronic phase after at least one cycle of standard chemotherapy and imatinib
  * Over 60 years of age with relapse within 6 months after completion of last chemotherapy
  * Over 60 years of age with blast count < 30% within 10 days before study entry
* Related HLA-haploidentical natural killer cell donor available
* No severe organ damage (by clinical or laboratory assessment)
* Performance status 50-100%
* No evidence of active infection on chest X-ray
* No active fungal infection

Exclusion Criteria:

* Active central nervous system (CNS) leukemia
* Pleural effusions large enough to be detectable by chest x-ray
* Pregnant or nursing (positive pregnancy test)
* Fertile patients must use effective contraception
* Less than 60 days since prior transplant
* Less than 3 days since prior prednisone
* Less than 3 days since other prior immunosuppressive medication

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bachanova V, Cooley S, Defor TE, Verneris MR, Zhang B, McKenna DH, Curtsinger J, Panoskaltsis-Mortari A, Lewis D, Hippen K, McGlave P, Weisdorf DJ, Blazar BR, Miller JS. Clearance of acute myeloid leukemia by haploidentical natural killer cells is improved using IL-2 diphtheria toxin fusion protein. Blood. 2014 Jun 19;123(25):3855-63. doi: 10.1182/blood-2013-10-532531. Epub 2014 Apr 9. PMID 24719405

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Relapsed/Refractory Acute Myeloid Leukemia: Patients who met study criteria - relapsed or refractory acute myelogenous leukemia - and were enrolled.
Period: Overall Study
Arm/Group | Patients With Relapsed/Refractory Acute Myeloid Leukemia
Started | 21
Completed | 20 (Evaluable patients - received adequate natural killer (NK) cells)
Not Completed | 1
Not completed — Did not receive adequate NK cells | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Relapsed/Refractory Acute Myeloid Leukemia
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 17
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Natural Killer (NK) Cell Expansion
Description: Evaluation of expansion of donor allogeneic natural killer (NK) cells at day 14 following infusion (>100 donor-derived NK cells per uL of patient blood detectable at day +14).
Time Frame: Study Day 14
Measure: Number; unit: Participants
Groups:
- Patients With Relapsed/Refractory AML - Evaluable Group: Patients who are evaluable; received adequate (dose of 1.5-8 x 10^7/kg natural killer (NK) cells 14 days after treatment with chemotherapy and allogeneic NK cell-enriched immune therapy.
Arm/Group | Patients With Relapsed/Refractory AML - Evaluable Group
Number analyzed (Participants) | 20
Participants | 2

2. Secondary Outcome: Number of Patients With Complete Remission
Description: Clinical response is determined by achievement of a complete remission (CR) as judged by morphological criteria (< 1% blasts in bone marrow with neutrophil recovery).
Time Frame: Day 28-35
Measure: Number; unit: Participant
Arm/Group | Patients With Relapsed/Refractory AML - Evaluable Group
Number analyzed (Participants) | 20
Participant | 2

3. Secondary Outcome: Median Time to Disease Relapse (Months)
Description: Follow-up continued every 3 months after the allogeneic natural killer (NK) cell infusion, unless they were transplanted, relapsed or had progressive disease. Time in months to relapse of disease is calculcated from 1st day of treatment with NK cells. Relapse occurs when leukemia is detected in bone marrow or blood.
Time Frame: From 1st Day of treatment until death or receipt of bone marrow transplant.
Population: Only 2 of 20 patients that received adequate Natural Killer Cells achieved complete remission, and were therefore evaluable for the time to relapse endpoint.
Measure: Median (Full Range); unit: Months
Groups:
- Patients Achieving Complete Remission - Responders: Patients who achieved complete remission (CR) as judged by morphological criteria; only these patients can be judged for time to relapse.
Arm/Group | Patients Achieving Complete Remission - Responders
Number analyzed (Participants) | 2
Months | 7.3 [3.5 to 11]

4. Secondary Outcome: Overall Survival Time of Patients With Complete Remission
Description: Median number of months patients were alive after NK cell infusion.
Time Frame: From Day 1 of Treatment until death or patient received bone marrow transplant.
Measure: Median (Full Range); unit: Months
Arm/Group | Patients Achieving Complete Remission - Responders
Number analyzed (Participants) | 2
Months | 13 [7 to 19]

5. Secondary Outcome: Number of Patients With Complete Remission and Natural Killer Cell Expansion
Description: Includes patients who had both a complete remission of disease and an expansion of natural killer cells.
Time Frame: Day 14
Population: Unable to evaluate due to low complete remission rate.
Arm/Group | Patients With Relapsed/Refractory AML - Evaluable Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Events were monitored from Day 1 of study through Day 60 post-natural killer cell infusion.
Description: All "other" adverse events that occurred were expected and not captured.
Arm/Group | Patients With Relapsed/Refractory Acute Myeloid Leukemia
Serious Adverse Events (participants affected / at risk) | 19/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Relapsed/Refractory Acute Myeloid Leukemia (N=21)
Death due to progressive disease (General disorders) | 14 (14) — unrelated to study
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (1) — central nervous system
Hemorrhage, lung (Blood and lymphatic system disorders) | 1 (1) — pulmonary/upper respiratory-lung
Infection (Infections and infestations) | 4 (4) — Meningitis x2, pneumonia, associated with lymphopenia
Leukoencephalopathy (Nervous system disorders) | 1 (1) — radiographic findings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes